CLINICAL TRIAL: NCT00655161
Title: A Pilot Phase 2 Trial of the Immunogenicity, and Safety of GI-4000; an Inactivated Recombinant Saccharomyces Cerevisiae Expressing Mutant Ras Protein, as Consolidation Therapy Following Curative Treatment for Stage I-III Non-Small Cell Lung Cancer (NSCLC) With Tumor Sequence Confirmation of K-ras Mutation
Brief Title: A Pilot Phase 2 Trial of the Immunogenicity, and Safety of GI-4000; an Inactivated Recombinant S. Cerevisiae Expressing Mutant Ras Protein, as Consolidation Therapy Following Curative Treatment for Stage I-III Non-Small Cell Lung Cancer (NSCLC) With Tumor Sequence Confirmation of K-ras Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlobeImmune (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GI-4000-03
Record Dates: First submitted 2008-04-02; First posted 2008-04-09 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: NSCLC
Keywords: NSCLC; Cancer Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: GI-4000 — subcutaneous injection, 40YU weekly for 3 weeks followed by monthly for 6 months them quarterly until recurrence

SUMMARY:
This is a consolidation therapy trial evaluating GI-4000 in subjects with NSCLC treated with curative intent who are disease free at their first post-treatment restaging assessment.

DETAILED DESCRIPTION:
NSCLC is the deadliest form of human cancer, killing approximately 150,000 people a year in the United States. The best treatment for NSCLC is surgical resection. For patients with inoperable or unresectable NSCLC chemotherapy and radiation is used as first line therapy. This is a consolidation therapy trial evaluating GI-4000 in subjects with NSCLC treated with curative intent who are disease free at their first post-treatment restaging assessment. These subjects must also have a ras mutation.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven stage I-III NSCLC
* Confirmed product related ras mutation
* ECOG performance status of less than or equal to 2
* greater than or equal to 18 years of age

Exclusion Criteria:

* History of a previous cancer
* History of splenectomy
* History of Crohns disease or ulcerative colitis
* History of major organ transplantation
* Concurrent or chronic steroid therapy
* History of allergy to yeast
* Presence of an unstable or poorly controlled medical condition
* Pregnant or nursing mothers
* Positive skin test to yeast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Immune response to GI-4000 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Chaft, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States